CLINICAL TRIAL: NCT02303925
Title: Feasibility of Superior Rectal Artery Embolization for the Treatment of Hemorrhoidal Disease
Acronym: EMBORRHOID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-41
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2016-08

CONDITIONS: Hemorrhoidal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- coils (Experimental)
  Interventions: Device: NESTER COILS

INTERVENTIONS:
Device: NESTER COILS

SUMMARY:
With an estimated prevalence between 4 and 35%, the hemorrhoidal disease is the most frequent proctologic disease. Its symptoms are mainly rectorrhagia, externalization of the hemorrhoidal cushions (muco-hemorrhoidal prolapse), and/or pain and pruritus. Its acute complications (external and/or internal thromboses) are unpredictable.

Surgical treatment concerns approximately 10% of patients with diagnosed hemorrhoidal pathologies. The elective ligature of the arteria haemorrhoidalis under trans-anal Doppler scanning was developed in order to reduce the postoperative morbidity of hemorrhoidal surgery. This technique consists in a ligation of the superior rectal artery under Doppler control in order to decrease the blood flow within the hemorrhoids and therefore to reduce them. It is effective in the treatment of internal hemorrhoidal pathology without prolapse (grade II). The complications rate is low and estimated between 2 and 12% : rectorrhagia (4.3%), thrombosed hemorrhoids (1,8%), fissure (0,8%), acute urine retention (0,7%).

With the major advances in interventional radiology such ligation could be performed by an endovascular coil embolization. Until now no direct study exists on the subject but several case reports show the feasibility of an embolization of the superior rectal arteries for rectorrhagia of various etiologies such as the hemorrhoidal disease.

Endovascular access should increase the selectivity of the embolization compared to the Doppler scanning technique. Indeed the arteriography makes it possible to scan all branches of the superior rectal artery and therefore to occlude permanently the branches that feed the hemorrhoidal plexuses. Moreover the endovascular embolization technique should avoid the main complications of the trans-anal access technique.

The primary objective of this study is : the assessment of the efficacy of endovascular coil embolization of the superior rectal arteries in the management of the symptoms of the hemorrhoidal disease grade II and III. The secondary objective is : the assessment of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from a symptomatic hemorrhoidal disease stage II or III (history of prior medical treatment or instrumental do not prohibit the inclusion in the study)
* Patient agreeing to participate in the study and who signed an informed consent
* Patient willing to lend to post-operative monitoring for a year
* Patient assured social

Exclusion Criteria:

* Diseases and colorectal proctologic / History proctologic
* Acute Complication hemorrhoidal disease course (thrombosis)
* History of proctology surgery for hemorrhoidal disease
* Anal stenosis congenital or acquired
* Chronic anal fissure, anal suppuration associated
* Chronic Inflammatory Bowel Disease
* History of colorectal cancer
* History of rectal resection and / or sigmoid
* Rectal prolapse
* Comorbidities
* Portal hypertension
* Severe atherosclerotic pathology (significant stenosis in aorto-iliac-femoral artery or branches for visceral).
* General Affection responsible for a disorder of hemostasis objective (hemophilia, von Willebrand disease thrombocytopenia) and anticoagulants.
* Psychiatric disorder making it impossible informed of and / or postoperative care
* Neurological disease directly or indirectly involving the rectosphinctérienne motor (multiple sclerosis, spinal cord injury or nerve root, polyneuropathy).
* Patients whose condition appears too insecure or taking steroids or immunosuppressive leading to an unacceptable surgical risk.
* Background
* Pregnancy declared (the existence of effective contraception will be checked for women of childbearing age)
* Major Trust
* Patients who do not speak French, refusing or unfit for monitoring proposed in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12-14 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Decrease of the felt pain | 26 MONTHS
  It will be expected a decrease of the felt pain at least of 2 points measured by visual analog scale for patients treated by coil embolization

SECONDARY OUTCOMES:
Reaaparition or obstinacy of the hemorroidal symptoms | 26 months
  Reaaparition or obstinacy of the symptoms will be assess by clinical exam at 1,3,6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille; vincent vidal, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France